CLINICAL TRIAL: NCT01159873
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending-Dose Study to Characterize the Safety, Pharmacokinetics, and Pharmacodynamics of CEP-37251 in Healthy Postmenopausal Women
Brief Title: Single Ascending-Dose Study to Characterize the Safety, Pharmacokinetics, and Pharmacodynamics of CEP-37251 in Healthy Postmenopausal Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been stopped by sponsor decision
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C37251/1080
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Bone Loss; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CEP-37251 (Experimental)
  Interventions: Drug: CEP-37251
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CEP-37251 — up to 5 subcutaneous (sc) doses (given sequentially in cohort groups) of CEP-37251 (0.03, 0.1, 0.3, 1.0, and 3.0 mg/kg) will be studied. After all 5 sc doses have been studied, an intravenous (iv) dose of 0.3 mg/kg will be studied.
  Arms: CEP-37251
Drug: Placebo — up to 5 subcutaneous (sc) doses (given sequentially in cohort groups) of Placebo (0.03, 0.1, 0.3, 1.0, and 3.0 mg/kg) will be studied. After all 5 sc doses have been studied, an intravenous (iv) placebo dose of 0.3 mg/kg will be studied.
  Arms: Placebo

SUMMARY:
Study to Characterize the Safety, Pharmacokinetics, and Pharmacodynamics of CEP-37251 in Healthy Postmenopausal Women.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a postmenopausal woman aged 40 years or greater but less than 75 years.
* The subject is ambulatory and healthy as judged by medical examination, medical history, and clinical chemistry, hematology and urinalysis at screening.
* The subject has a body weight greater than 50 kg but no more than 100 kg with a body mass index (BMI) of 18 to 35 kg/m2).
* The subject has a normal or clinically acceptable ECG.
* The subject is willing to give written informed consent prior to any study-related procedures being conducted.
* The subject is willing and able to comply with the study restrictions and to remain in the study center for the required inpatient period.

Exclusion Criteria:

* The subject has received any of the following medications within the 6 months prior to enrollment:

  * hormone replacement therapy
  * selective estrogen receptor modulator (SERM) therapy such as raloxifene
  * elemental calcium supplementation >1.5 g/day
  * Vitamin D supplementation >1000 IU per day
  * calcitriol or other Vitamin D analogs (eg, alfacalcidol, doxercalciferol, or paricalcitol)
  * calcitonin or parathyroid hormone
  * chronic use of glucocorticoids NOTE: Acute use of glucocorticoids may be permitted after consultation with the medical monitor if it occurred a minimum of 6 weeks prior to enrollment
  * anabolic steroids
* The subject has received bisphosphonates or fluoride within the 12 months prior to enrollment.
* The subject has any of the following concomitant conditions:

  * hypo- or hyperthyroidism. NOTE: Subjects with treated hypothyroidism with normal thyroid parameters may be allowed to participate in the study at the discretion of the investigator and medical monitor.
  * hypo- or hyperparathyroidism
  * recent fracture (within 6 months)
  * osteomalacia, Paget's Disease, osteopetrosis, osteogenesis imperfect, or other bone disease
  * rheumatoid arthritis or psoriatic arthritis
  * acute osteoarthritis or gout
  * chronic kidney disease or renal failure defined as an eGFR (by MDRD equation) 30 mL/min/1.73 m2 or less
* The subject is receiving immunosuppressant drugs.
* The subject is currently participating in another investigational study or has received any investigational drug within 60 days before the dose of study drug.
* The subject has evidence of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, psychiatric, or cerebral disease, or malabsorption syndrome.
* The subject has a known history or evidence of malignancy, lymphoproliferative, or neoplastic disease with the exception of being successfully treated for basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia.
* The subject has had any substantial change in levels of physical activity or participated in intense physical activity (e.g., marathon training) within the 6 months prior to the dose of study drug.
* The subject has any other clinically significant disease or disorder or factors, such as substance abuse, which in the opinion of the investigator, make the subject ineligible for participation in this study.
* The subject has a known or suspected hypersensitivity or idiosyncratic reaction to any compound present in the study drug or placebo.
* The subject has habitually consumed, within the past 2 years, more than 21 units of alcohol per week, or has a history of alcohol, narcotic, or any other substance abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR). NOTE: A unit of alcohol is equal to approximately 30 ml of spirits, 100 ml of wine, or 260 ml of full-strength beer.
* The subject has, within 2 weeks before administration of the dose of study drug, a clinically significant excessive consumption of coffee, tea, and/or other caffeine-containing beverage or food (i.e., 600 mg of caffeine or more per day, or 5 or more cups of coffee per day), or a combination of any of these beverages or foods.
* The subject has had, within 4 weeks before the dose of study drug, a clinically significant illness or, within 1 week before the dose of study drug, has had any acute illness, or at screening or on the day before the dose of study drug, has symptoms of any clinically significant or acute illness.
* The subject has, after resting for 5 minutes, elevated blood pressure (defined as a systolic blood pressure of more than 140 mm Hg for subjects ≤50 years of age or 155 mm Hg for subjects >50 years of age and/or a diastolic blood pressure of more than 90 mm Hg) or has low blood pressure (defined as systolic blood pressure of less than 90 mm Hg and/or diastolic blood pressure of less than 45 mm Hg).
* The subject has, after resting for 5 minutes, a pulse less than 45 beats per minute (bpm). The subject has, after resting for 5 minutes, a pulse more than 90 bpm for subjects ≤50 years of age or a pulse more than 100 bpm for subjects >50 years of age.
* The subject has a positive test result for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C or human immunodeficiency virus (HIV).
* History of any clinically important drug and/or vaccine allergies.
* The subject has received immunization with a live or live attenuated vaccine within 3 months prior to the dose of study drug or has immunization with a live or live attenuated vaccine planned within 3 months after the dose of study drug.
* The subject has an ongoing active systemic infection requiring treatment or a history of severe infection, such as hepatitis or pneumonia, in the 3 months prior to the dose of study drug. Less severe infections in the 3 months prior to the dose of study drug are permitted at the discretion of the investigator and medical monitor.
* The subject has a positive alcohol serum, urine, or breath test result or a positive urine drug screen (UDS).

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Characterize the Overall Safety Assessment of CEP-37251 | 70 days
  Measurements include adverse events, laboratory results, vital sign measurements, electrocardiogram findings, physical examination findings, injection site evaluations, concomitant medication usage, immunophenotyping test results, and immunogenicity test results.

SECONDARY OUTCOMES:
Characterize the Overall Pharmacokinetic Profile of CEP-37251 | 70 days
  Pharmacokinetic parameters include Cmax (Maximum Concentration) and AUC (Area Under the Curve) plasma concentration
Characterize the Overall Pharmacodynamic Effect of CEP-37251 | 70 days
  Pharmacodynamic effect as measured by markers of bone metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Clinical Pharmacology and Experimental Medicine, MD, Study Director — Cephalon
Locations (1):
- Cephalon Investigational Site, Adelaide, Australia